A randomized, placebo-controlled, double-blinded trial of the safety and efficacy of tecovirimat for the treatment of adult and pediatric patients with monkeypox virus disease

**PALM 007 Study Extension** 

15 April 2025

NCT06721585

# RESEARCH PARTICIPANT INFORMED CONSENT AND PRIVACY AUTHORIZATION FORM

**Protocol Title:** PALM 007: A randomized, placebo-controlled, double-blinded

trial of the safety and efficacy of tecovirimat for the treatment of adult and pediatric patients with monkeypox virus disease

**Sponsors:** United States National Institute of Allergy and Infectious

Diseases (NIAID), National Institutes of Health (NIH)

Democratic Republic of the Congo (DRC) Institut National de la

Recherche Biomédicale (INRB)

Principal Investigators: Jean-Jacques Muyembe-Tamfum, MD, PhD

Placide Mbala-Kingebeni, MD, PhD

Site: DRC, Central Africa

**Extension phase consent (SOC only)** 

#### **KEY INFORMATION**

This consent form describes a clinical research study and is designed to help you decide if you would like to be a part of the study. A clinical research study helps doctors test new ways to treat a disease or helps us collect information about how a disease affects people so we can learn more about it and possible future treatments.

This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. More information that may help you make a decision can be found in other sections of the document.

### What you should know about this study:

- You are being asked to join this clinical research study because you have severe monkeypox virus disease, which is also called mpox.
- You can take as much time as you need to review this form and discuss your study participation with your family, friends, and community as you feel comfortable and appropriate, in order to decide whether or not you would like to participate.
- Ask the study team to explain any words or information that you do not understand.
- You are a volunteer and you do not have to join this study.
- Your other option is to continue receiving any other care you have already been receiving, which would include the standard of care treatment for mpox.
- If you join the study, you can change your mind later. You can decide not to take part or you can quit at any time. There will be no penalty or loss of benefits if you decide not to join or to quit the study. Your care within your community will not be affected.
- During the study, we will tell you if we learn any new information that might affect whether you wish to continue to be in the study.
- If you are signing for a person who cannot consent for themselves, such as a child or a person who is too sick to read and understand this, the word "you" in this consent form refers to that person.

• If you decide to participate in this study, you will review this document with a member of the study staff and will be requested to sign and date at the end of this form to show that your questions have been answered and that you want to take part in the study. A copy of this signed/marked informed consent will be provided to you. This consent must be signed/marked before any study procedures are performed.

### What is this study about?

We are looking for new treatments for mpox disease, which is caused by infection with the monkeypox virus. Mpox can make people very sick and some people can die from it. There are no medicines approved in Africa to treat mpox. There is one drug approved in Europe to treat mpox, but it has not been used in many people with the disease.

In the first part of this study, we collected more information about how well this drug works to treat mpox. The results from that part of the study showed that the drug we tested, called tecovirimat (TPOXX), did not help treat mpox. However, we plan to continue to treat people with mpox using standard care under this study so we can keep learning more about mpox disease. So on this part of the study, we are only giving the standard of care treatment for mpox.

### What will happen on this study that is different than if you were not on this study?

If you join this study, you will need to be in the hospital until you recover from mpox. You will be able to leave the hospital when you have recovered from mpox. While you are in the hospital, you will receive standard care for mpox. For the research, we need to collect more information on your health and get more frequent blood samples than you would have if you were not in this study. We will test these samples to figure out when you have recovered from mpox. We may ask for biopsy samples from your mpox lesions. After that, we will examine the lesions every day until they have healed. We will take a swab sample from your eye if you have eye symptoms or lesions touching your eye.

After you have recovered from mpox and leave the hospital, if you get new mpox symptoms, you can come back for a sick visit. We will collect information about your health, take more blood samples, count your new lesions, and take swab samples from your lesions and your eye if you have eye symptoms or lesions touching your eye. We will also offer you standard treatment.

If you deliver a baby or have a miscarriage, we may take a swab of fetal skin lesions, products of conception, placenta, amniotic fluid, and umbilical cord to look for the monkeypox virus. If you have a miscarriage or a baby, we may ask you information about this even if you have already finished your participation in this study.

Your total amount of time on this study will be 59 days. If you do not come back for a sick visit during this time period, you will not have any more visits for this study. You will be compensated for the time and inconvenience of taking part in the study.

### What are the main study risks?

When we collect blood for our research, even though we may collect more blood than is normally taken, it will be done the usual way and the risks do not differ in this study from when you normally get blood drawn.

If we take biopsy samples from your mpox lesions, you may have some pain or burning when we inject the numbing medicine into your skin before taking the biopsy. The numbing medicine may also irritate the skin, or rarely cause an allergic reaction, which can be treated with medicine. There may be minor bleeding or redness near the biopsy site, and the biopsy will leave a scar. There is a small chance of an infection at the biopsy site, which may need to be treated with antibiotics.

#### Are there benefits to being in the study?

You will receive the regular medical care for mpox. You will have frequent testing on this study that can give your doctors more details about your health. The study staff will follow your health closely while you are on this study.

The rest of this document will describe more about the research study. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document.

# 1. What will happen if you want to join this study?

If you think you may want to join this study, we will describe the study and answer any questions you may have. You can also talk to your friends and family about the study.

If you agree to be in the study, we will ask you to sign this consent form. When you sign your name or put your mark on the consent form, it means that you agree to be in the study. You can change your mind at any time and leave the study. If you decide not to join the study or to leave the study later, you will not lose any regular health care services you already are getting. About 600 people were included in the first part of this study. We plan to enroll about 400 in this part of the study.

### 2. What does the study involve?

If you decide to join this study, you will stay at the hospital for treatment of your mpox. While you are in the hospital, you will get the supportive care that you would typically get for mpox. We will measure your height and weight, and we will measure the size of the upper arm for children who are 3 months to 5 years old. We will also take vital signs, check your health, and review your mpox symptoms frequently while you are in the hospital. We may also request the results of tests you have done as part of your medical care to review as part of this study. We will collect 1-2 tbs of blood every few days until discharge. We will take a swab sample from your eye if you have eye symptoms or lesions touching your eye. We will use these samples to monitor your health, see how your body responds to the standard treatment, and to test for the monkeypox virus. We may also test your blood for malaria. If you agree, we will test your blood for HIV (the virus that causes AIDS). This test may not be done until later, so we may not have a result to give you right away. A member of the study team will explain this test further. If you do not want your blood to be tested for HIV, you are still able to participate in this study. According to DRC guidelines, the study team will provide you HIV test counseling. If you have a positive test, meaning that you have HIV infection, the study staff/counselor or an official from the Health zone will attempt to contact you to tell you what that means and will refer you for treatment according to the national guidelines, as the treatment for HIV will not be provided as

part of this study. The study team may also report positive results to the necessary authorities according to the guidelines of DRC.

While you are in the hospital, we may ask for biopsy samples from your mpox lesions. You can say no to this and still be in the study. If you agree, we will first numb the area by injecting a numbing medicine under the skin. At least one tissue sample up to 8 mm in size will be removed using a small, sharp instrument (skin punch) or scalpel depending on skin thickness. Biopsy sites will be closed with stiches if needed. The stiches will dissolve, so you do not need to come back to have them removed.

You will be allowed to go home once all of your mpox skin lesions have healed and a blood test shows that you no longer have monkeypox virus.

If you get new mpox symptoms after you leave the hospital, you may come back for a sick visit. We will take more blood samples, count your new lesions, and take swab samples of your lesions. If you have any eye symptoms or lesions touching your eyelids, we will also take a swab from your eye. We will use the samples to check your health and to test for the monkeypox virus. We will also offer you standard treatment. You will be done with this study after 59 days.

If you deliver a baby or have a miscarriage, we may take a swab of fetal skin lesions, products of conception, placenta, amniotic fluid, and umbilical cord to look for the monkeypox virus. If you have a miscarriage or a baby, we may ask you information about this even if you have already finished your participation in this study.

As part of this study, we will do some routine medical tests on your samples. We will share the results of these tests with you, and your health information will go in your medical record. We will also store and use some of your samples for research tests, and you will not receive these results.

# 3. What are the other risks or discomforts of the study?

We will insert a new, clean needle into a vein in your arm to take blood. You may feel a pinch when the needle goes through your skin. A bruise may appear where it was put in. You may also have swelling and redness, and the area may be sore. These things are common and should go away in a couple of days. Some people faint when they have blood drawn. There is a very small chance of an infection where the needle goes into your vein. An infection could be treated with antibiotics.

If you have a skin biopsy, you may have some pain or burning when the numbing medicine is injected under your skin. It may also irritate the skin, or rarely cause an allergic reaction, which can be treated with medicine. There may be minor bleeding or redness near the biopsy site. A skin biopsy will leave a scar at the site. There is a very slight chance that the scar will become raised and hard. Very rarely, the biopsy site might get infected. Signs of an infection include growing redness, warmth, swelling, pain, or irritation around the cut. Please contact us if you have any problems on your skin where the biopsies were done, like scars that bother you or an infection. We can refer you for treatment or give you antibiotics if needed.

Collection of the swab samples may be uncomfortable, but should not hurt.

We will be careful to keep your study information confidential, but there is a small risk that someone not involved in the study could get this information.

### 4. Are there benefits to being in the study?

You will receive the regular medical care for mpox. You will have frequent testing on this study that can give your doctors more details about your health. The study staff will follow your health closely while you are on this study.

Your participation in this study is important to learn more about how to treat mpox. It will help in the development of treatments for mpox and may in the future help people all over the world.

# 5. What will happen to your samples and personal information?

We will store your samples and data (information) for a very long time to use for future research on mpox or other similar types of diseases after this study is over. This is in addition to them being used and stored for research testing under this current study. Your samples will be stored in a secure location, and your data will be placed in a secure electronic system. Your stored samples and data will be marked with a code and not with your name. Only researchers linked to this study can get the codes.

In addition to our own use, we may share your samples and data with other researchers for future research with or without information that could identify you. If we include information that could identify you, we must get approval from the DRC ethics board. Other information, such as your sex, age, or health history might also be shared. Results from future research will not be shared with you. Your samples will not be sold. You will not be paid for any products that result from this research.

The only risk of allowing us to store your samples would be an accidental release of your identity.

| 0 1 | ion for my samples and data to be stored and ve (please check one option below): | dused for future studies as |
|---|---|---|
| Yes | | |
| No | | |

In addition, we might remove any information from your specimens and data that could identify you, and then share them with other researchers for future studies. If we do this, there will be no way to know that they came from you. We would not be able to remove your specimens or data from these studies or prevent their use in future studies because we would not be able to tell which specimens or data belong to you. We want to make sure that you understand that this is a possibility if you participate in this study.

If you agree to the storage of your samples and data now but you change your mind later and decide you do not want us to store your samples or data, please let us know.

We will do our best to follow your wishes but cannot promise that we will always be able to destroy your samples or data.

### 6. Will it cost you anything to be in this study?

It will not cost you anything to be in this study. Hospitalization and standard care will be given for free to everyone participating in this study. You and 1 person who are with you will receive meals each day that you are in the hospital.

## 7. Will you be paid if you join this study?

You will be compensated for your time and inconvenience as follows.

A stipend of US\$4 in CDF will be provided daily to you and one person who is with you during the hospitalization period.

Travel will be provided for you and one person who accompanies you to and from a sick visit.

## 8. Who is watching over this study?

In addition to the investigators and sponsors who are overseeing this study, the DRC ethics board will also be watching over this study and has the authority to stop it at any time.

# 9. How will your privacy be protected?

We will keep your study information private. All files with information that could identify you will be kept in locked cabinets or secure computers. People responsible for making sure that the research is done properly may look at your study records. This might include people from the DRC and the US including the NIH and their designees. All of these people will also keep your identity private. Results from this study, but not your identity, may be shared with other researchers, local medical providers, or government health organizations to help them better understand monkeypox virus infection and treatment.

# 10. Could you be removed from the study early?

You could be taken out of the study early if you do not or cannot follow the study requirements, if the study doctors feel it is better for you to be removed from the study, or if the study is stopped early. If you are removed from the study early, we will still use your stored samples and data for research unless you ask us not to.

# 11. What if the researchers learn new information during this study?

Results of this study or other scientific research may affect your willingness to continue to take part in this study. During the course of the study, you will be informed of any significant new findings (either good or bad), such as changes in the risks or benefits resulting from participation in the research or new alternatives to participation that might cause you to change your mind about continuing in the study. If new information is provided to you, your consent to continue participating in this study will be re-obtained.

# 12. What other things should you know about this research study?

### a. ClinicalTrials.gov

A description of this study is on the internet at http://www.ClinicalTrials.gov. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **b.** Conflict of Interest

Any potential conflict of interest will be resolved according to the guidelines of the local ethics review committee of DRC.

### c. What is the Ethical Review Committee and how does it protect you?

Your government's ethics committee will review this study. It protects the rights and welfare of the people taking part in research studies. You can contact Paul Samson Lusamba Dikassa, President of the Kinshasa School of Public Health ethics committee (KSPH EC) (Tel: +243975012791) or Mbongo Pasi Moke Sangol, Vice-President of the KSPH EC in DRC (Tel: +243817493194) to answer questions you may have about being part of this study and your rights as someone who is in a study.

#### d. What do you do if you have questions about the study?

If you have questions about the study, you may contact the principal investigators. Prof. Jean-Jacques Muyembe-Tamfum can be reached by phone: +243 892625954, or by email: jjmuyembet@gmail.com. Dr. Placide Mbala-Kingebeni can be reached by phone: +243 822851584, or by email: mbalaplacide@gmail.com.

e. What should you do if you are injured or ill as a result of being in this study? We do not expect any harm from participating in this study. However, unforeseeable risks may be present. The study doctors will give you short-term medical care if you are hurt by being in this study.

| If you agree to be in this study, please sign or put your fingerprint below. | | | | | | | |
|---|---|---|---|---|---|---|---|
| Signature or fingerprint of participant or guardian | Date: | dd | _/_<br> | <u>/</u><br>m : | уу | Time: | |
| Printed name of participant or guardian | | | | | | | |
| Signature of investigator/designee | | | | Date: | dd | //<br> | /yy |
| Printed name of investigator/designee | | | | | | | |

| Complete if participant is illiterate: | |
|---|---|
| Witness to Consent | Interview |
| On the date given next to my signature, I witnessed study named above in this document. I attest that the explained to the subject, and the subject indicated the adequately addressed. | e information in this consent form was |
| Signature of witness | Date://<br>dd mm yy |
| Printed name of witness | |